CLINICAL TRIAL: NCT00722722
Title: The Impact of Velcade(TM)on Antibody Secreting Cells in Sensitized Renal Allograft Candidates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Stegall, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-000556
Record Dates: First submitted 2008-07-23; First posted 2008-07-28 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 dose group (Active Comparator): 4 doses of bortezomib (1.3mg/m^2 of body surface area)
  Interventions: Drug: Bortezomib
- 16 dose group (Active Comparator): 16 doses of bortezomib (1.3mg/m^2 of body surface area)
  Interventions: Drug: Bortezomib
- 32 dose group (Active Comparator): 32 doses of bortezomib (1.3mg/m^2 of body surface area)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Velcade given in four-dose cycles intravenously (through a vein).
  Other Names: Velcade(TM)

SUMMARY:
Patients planning to have kidney transplantation who are sensitized to their donors have high levels of donor specific alloantibodies. High levels of donor specific antibodies put kidney transplant recipients at risk for rejection very early after transplant. This study is trying to determine if the drug bortezomib (Velcade ™) can reduce donor specific alloantibodies to a level that permits kidney transplantation without a high risk for rejection.

DETAILED DESCRIPTION:
The study is designed to assess the impact of in vivo treatment of bortezomib on anti-human leukocyte antigen (HLA) production by normal antibody secreting cells (ASC) in sensitized renal allograft candidates. The design involves treatment of subjects with bortezomib using one of three dosing regimens (4 doses, 16 doses or 32 doses of bortezomib). Using novel assays, anti-HLA production is determined by measuring the bone marrow derived ASC at baseline (prior to therapy) and after treatment (at day 14, 3 days after the last bortezomib dose). Paired data are used with patients serving as their own controls. Finally, the safety of bortezomib is evaluated by monitoring total serum antibody levels and the incidence of side effects (primarily neuropathy) at 1 month, the final follow-up point.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

  * Female subject is post-menopausal, surgically sterilized, or she and/or sexual partner are willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
  * Male subject agrees to use an acceptable method for contraception for the duration of the study.
  * Renal transplant candidates who otherwise meet our acceptance criteria.
  * Evidence of alloantibody in their serum (panel reactive antibody >20% and specificities determined by single antigen flow bead assay).
  * Sensitized patients with no living donors or have donor-specific antibody levels too high to undergo successful transplantation using our current protocols (T or B cell crossmatch channel shift >500).

Exclusion Criteria:

* Patient has a platelet count of <30 x 10^9/L within 14 days before enrollment.

  * Patient has an absolute neutrophil count (ANC) of <1.0 x 10^9/L within 14 days before enrollment.
  * Patient has >Grade 2 peripheral neuropathy within 14 days before enrollment.
  * Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator as not medically relevant.
  * Patient has hypersensitivity to bortezomib, boron or mannitol.
  * Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
  * Patient has received other investigational drugs within14 days before enrollment.
  * Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
  * Diagnosed or treated for malignancy within 5 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
  * Contraindication to kidney transplantation-active infection, comorbid medical conditions, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Diwan TS, Raghavaiah S, Burns JM, Kremers WK, Gloor JM, Stegall MD. The impact of proteasome inhibition on alloantibody-producing plasma cells in vivo. Transplantation. 2011 Mar 15;91(5):536-41. doi: 10.1097/TP.0b013e3182081333. PMID 21283064
- [Derived] Moreno Gonzales MA, Gandhi MJ, Schinstock CA, Moore NA, Smith BH, Braaten NY, Stegall MD. 32 Doses of Bortezomib for Desensitization Is Not Well Tolerated and Is Associated With Only Modest Reductions in Anti-HLA Antibody. Transplantation. 2017 Jun;101(6):1222-1227. doi: 10.1097/TP.0000000000001330. PMID 27379560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 Dose Group | 16 Dose Group | 32 Dose Group
Started | 3 | 5 | 10
Completed | 3 | 5 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Dose Group | 16 Dose Group | 32 Dose Group | Total
Number analyzed (Participants) | 3 | 5 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (3.5) | 40.4 (11.4) | 39.5 (6.6) | 39.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7 | 14
  Male | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Response to Bortezomib Monotherapy
Description: Response to treatment with Bortezomib (BTZ) alone was defined as a reduction in serum Donor Specific Alloantibody (DSA) levels following treatment. DSA levels were measured prior to treatment and after treatment. A good response occurred if all DSA were reduced. A partial response when a reduction was observed in at least one DSA, but not all DSA. No response occurred when no reduction of any DSA was attained.
Time Frame: 6 months
Population: In the 32 dose group, one patient received a kidney transplant with a B-cell flow cytometric crossmatch channel shift of less than 300 after dose 20 and was transplanted with a positive crossmatch donor. This patient was then excluded from further DSA analysis.
Measure: Number; unit: participants
Arm/Group | 4 Dose Group | 16 Dose Group | 32 Dose Group
Number analyzed (Participants) | 3 | 5 | 9
participants
  Good Response | 0 | 0 | 0
  Partial Response | 1 | 1 | 6
  No Response | 2 | 4 | 3

ADVERSE EVENTS:
Time Frame: Subjects were followed for 6 months. Before each drug dose, subjects were evaluated for possible toxicities that may have occurred after the previous doses(s).
Arm/Group | 4 Dose Group | 16 Dose Group | 32 Dose Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 Dose Group (N=3) | 16 Dose Group (N=5) | 32 Dose Group (N=10)
Anemia Grade 1 (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 4 (4)
Anemia Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 6 (6)
Thrombocytopenia Grade 1 (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 7 (7)
Thrombocytopenia Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea/Vomiting Grade 1 (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5)
Diarrhea Grade 1 (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Diarrhea Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Flu-like symptoms Grade 1 (General disorders) | 0 (0) | 2 (2) | 6 (6)
Myalgias Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 7 (7)
Chills Grade 1 (General disorders) | 0 (0) | 0 (0) | 5 (5)
Fatigue Grade 1 (General disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue Grade 2 (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes